CLINICAL TRIAL: NCT03104504
Title: A System of Safety: Preventing Suicided Through Healthcare System Transformation
Brief Title: A System of Safety (SOS)
Acronym: SOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Edwin Boudreaux, Vice Chair, Director of Research, University of Massachusetts, Worcester
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: H00011407; 1R01MH112138-01 (NIH)
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Suicide
Keywords: Suicide Screening; Safety Planning
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Design
Who Masked: Participant
Masking Description: This was an implementation study that implemented various suicide related best practices into routine care. Data for patients who presented for care were included in the respective phase of the study based on the location and date of presentation. They were not aware they were in a study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention (No Intervention): Baseline Retrospective Chart Reviews that are conducted on subjects for the one year period prior to the implementation of the study will serve as the control.
- Intervention (Other): The intervention targets will be the following suicide-related clinician behaviors.
  * suicide risk screening
  * safety planning
  * means restriction counseling
  * Post-acute care follow-up calls A Lean Implementation Strategy: The Implementation of the intervention targets guided by Lean; is expected to increase suicide-related clinician behaviors
  Interventions: Behavioral: Suicide Risk Screening; Behavioral: Safety Planning; Behavioral: Care transition facilitation; Behavioral: A Lean Implementation Strategy

INTERVENTIONS:
Behavioral: Suicide Risk Screening — Suicide risk screening will be implemented as the standard of care for all patients who present for treatment.
  Arms: Intervention
Behavioral: Safety Planning — Suicide screen-positive patients who are to be discharged from the hospital will receive personalized safety planning by a mental health clinician or nurse that includes means restriction counseling as a step in the safety plan.
  Arms: Intervention
Behavioral: Care transition facilitation — Include post-acute telephone phone call follow-up to foster engagement with outpatient care and problem solving within 24 hours of discharge
  Arms: Intervention
Behavioral: A Lean Implementation Strategy — The Interventions will be implemented using Lean performance improvement strategies
  Arms: Intervention

SUMMARY:
SOS will identify evidence based best practices consistent with Zero Suicide's six specific recommended clinical actions (A.2.) and use them to develop standardized clinical protocols for each care setting, clinical unit, population serviced, and clinical discipline. Using Lean CQI, the investigators will tailor, implement, and improve adherence to these protocols. To support feasibility, SOS will use a phased roll out and a hub-and-spoke design. The intervention targets will be suicide-related clinician behaviors. The investigators will aspire to adopt best practices and measure all six recommended performance elements; however, for feasibility, the research evaluation will focus on suicide risk screening, safety planning, means restriction counseling, and post-acute care follow-up calls. The primary patient outcomes will be suicide risk identification, suicide, suicide attempts, and suicide-related emergencies requiring acute care. The investigators will examine potential mechanisms of action and moderators, and conduct a cost effectiveness analysis of SOS versus usual care. The investigators will employ a stepped wedge design and follow individuals for 6 to 54 months. Outcomes, clinician behaviors, and other variables will be gathered through: (1) EHR data extraction, (2) claims data from UMMHC and the MA All Payer Claims Database, (3) random medical chart abstractions, (4) MA state vital statistics and National Death Index (NDI), (5) clinician surveys, (6) Lean evaluations and process observations, and (7) patient fidelity interviews. Data will be analyzed using generalized linear mixed models.

DETAILED DESCRIPTION:
The System of Safety (SOS) project will catalyze and expand the investigators existing efforts to transform suicide risk detection and suicide prevention across the UMass Memorial HealthCare system (UMMHC), the largest healthcare system in central Massachusetts representing a catchment area of 1.06 million people. This effort will span emergency department, inpatient, and primary care settings; engage medical and behavioral health clinicians; target adults and children; and support integration and collaboration across the entire system to provide a 360-degree safety net for patients at risk for suicide. Building on our previous and ongoing work, Zero Suicide's Seven Essential Elements of Care (Essential Elements) will be the foundation for an innovative continuous performance improvement (CQI) hub-and-spoke model whereby a central System Hub will work with Local Hubs and Spokes representing each setting and clinical unit. SOS will evolve over three phases. Phase 1 (months 1 - 12) will start with the emergency departments across the four UMMHC hospitals; Phase 2 (months 13 - 30) will extend the efforts to the inpatient medical and psychiatric units; and, Phase 3 (months 31 - 48) will expand to primary care settings. Overall, 39 clinical units will be engaged.

Consistent with central CQI tenets and the Zero Suicide model, the investigators will create protocols using best-practice approaches to identifying, assessing, managing, and intervening with suicidal patients while tailoring the approach to the particular clinical unit's unique needs and population. Units will learn from one another through regular collaborative work sessions, retreats, and cross departmental sentinel case reviews of suicides and suicide attempts. Fidelity to key components of the protocols will be measured.

The investigators will use a stepped wedge design with cluster randomization of clinical units, stratified by setting. Within each setting (Phase), the study population will consist of all patients seen in any of the clinical units during the pre-specified observation period before (Control) or after (Intervention) the unit's implementation start date. The investigators will follow these estimated 310,000 patients from their 1st encounter with a clinical unit through 6 months after Phase 3 ends (month 54). The investigators Aims assess the effect of SOS on its intervention targets (clinician behaviors) and on patient outcomes, using a system-level analytic strategy. The Specific Aims are:

Aim 1: Examine the impact of the SOS intervention on clinician-administered, standardized suicide risk screening and suicide risk identification across settings and clinical units.

H1: Likelihood of clinician-administered standardized suicide risk screening (an intervention target) at the time when a patient enters the study will increase monotonically with time since study initiation.

H2: Likelihood of suicide risk identification (patient outcome) at the time when a patient enters the study will increase monotonically with time since study initiation.

H3: The increasing likelihoods of screening and identification are attributable to SOS implementation.

Aim 2: Examine the impact of SOS on suicide related outcomes across settings and clinical units.

H4: As SOS is implemented across more settings and clinical units, the likelihood of receiving a best practice suicide prevention intervention by a clinician (intervention target) will increase among newly identified at-risk patients. This includes, but is not limited to, collaborative safety planning, means restriction counseling, and a post-acute care follow-up telephone call within 24 hours of discharge.

H5: SOS implementation will decrease the likelihood of suicide, suicide attempt, or suicide-related emergency requiring acute medical attention (patient outcomes) among newly identified at-risk patients.

H6: "Dose" of exposure to SOS will mediate the effect of SOS noted in H5.

Exploratory Aims: The investigators will also evaluate SOS from different perspectives by:

A: Exploring potential moderating and mediating factors, and potential mechanisms of action, such as:

EH1: Supportive organizational characteristics (e.g., embedded behavioral services on site, providing regular clinician-level performance feedback) will promote higher adherence to SOS implementation.

B: Exploring the population level effect of SOS on a subgroup of UMMHC patients that constitutes an Accountable Care Organization (ACO). For example, the investigators hypothesize that:

EH2: Suicide-related outcomes measured at the entire ACO population level (not just those encountering a clinical unit during the study period) will decrease monotonically during the study period (3-month increments).

C: Exploring the cost-effectiveness of the SOS intervention compared to usual care. The investigators hypothesize that EH3: The cost of SOS will be < $50,000/ quality-adjusted life year saved, a commonly used threshold.

ELIGIBILITY:
Inclusion Criteria:

* • Patients >12 years old

Exclusion Criteria:

* • Patients <12 years old

  * Adults unable to consent
  * Prisoners

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 493756 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Standardized suicide risk screening | 6 months after the Index ED Visit
  A completed suicide screen will be defined as any chart documentation of the presence OR absence of suicidal ideation AND presence or absence of a past suicide attempt (0=None documented, 1=Partial (+/- ideation OR attempt noted), 2=Complete (+/- ideation AND attempt noted).
Safety planning | 6 months after the Index ED Visit
  A safety plan will be defined as a written document collaboratively developed with the patient identifying steps to take when feeling suicidal. We will code it as 0=None, no documentation of a safety plan, 1=Partial (e.g., some steps but not all completed), or 2=Complete (all six steps completed).
Means restriction counseling | 6 months after the Index ED Visit
  a step in the Safety Plan Intervention includes means restriction counseling. We will code it as 0=None, no documentation of means restriction counseling, 1=Complete, documentation of means restriction counseling.
Care transition facilitation | 6 months after the Index ED Visit
  Include post-acute telephone phone call follow-up to foster engagement with outpatient care and problem solving within 24 hours of discharge (0 = Not completed, 1 = Completed).
Suicide risk identification | 6 months after the Index ED Visit
  A positive screen (i.e., identification) will be defined as patient endorsement of active ideation OR report of a lifetime suicide attempt. We will also examine ICD-10 codes assigned to each visit within claims data.
Suicide outcomes | 6 months after the Index ED Visit
  Suicide will be ascertained through MA vital statistics review with the DPH Suicide Prevention Program. We will match definite and suspected suicides against the study population. Suicide attempt will be defined as an ED visit or a hospitalization with: an ICD-10 code (i.e., intentional self-injury) OR Positive suicide attempt on an encounter day per the EHR templated screener. Suicide-related acute healthcare encounter will be defined as a suicide attempt (same criteria as above) OR a ICD-10 code (i.e., suicidal ideation) OR positive screen for suicidal ideation per the EHR templated screener

CONTACTS AND LOCATIONS:
Overall Officials: Edwin D Boudreaux, PhD, Principal Investigator — University of Massachusetts, Worcester; Catarina Kiefe, MD, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Memorial Health Care, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified database from this study, along with associated database documentation (see below), will be made available online three years after the dataset is closed, without cost to researchers and analysts. NIMH will host the dataset on the NIMH Limited Access Dataset website; access and use will be governed by its policies, which can be found at: http://www.nimh.nih.gov/health/trials/datasets/nimh-policy-for-distribution-of-data.shtml.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be become available in years, length to be determined.
Access Criteria: See plan description